CLINICAL TRIAL: NCT00646152
Title: A Phase I Double-Blind, Placebo-Controlled, Dose-Escalating Study to Evaluate the Safety and Tolerability of Topical Nasal Poly-ICLC
Brief Title: Poly-ICLC to Prevent Respiratory Viral Infections A Safety Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: 080093; 08-I-0093
Record Dates: First submitted 2008-03-27; First posted 2008-03-28 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2014-07-01

CONDITIONS: Influenza; Severe Acute Respiratory Distress Syndrome; Smallpox; Ebola; Unknown Respiratory Viruses
Keywords: Antiviral; Influenza; Interferon; Prophylaxis; SARS; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza, Human; Respiratory Distress Syndrome; Smallpox; Hemorrhagic Fever, Ebola | interventions — poly ICLC

INTERVENTIONS:
Drug: Poly-ICLC

SUMMARY:
This study will examine the safety of an experimental medication called Poly-ICLC, developed for preventing or reducing the severity of infections from influenza and other viruses acquired through the nose, mouth and lungs. The study is divided into two parts, in which Poly-ICLC is tested at different dose levels.

Healthy people between 18 and 70 years of age who have no chronic medical problems may be eligible for this study. Participants undergo the following procedures:

Part I

* Up to 7 days before Poly-ICLC administration: Medical history, physical examination and blood tests.
* Day 1: Nasal wash and Poly-ICLC administration. A small amount of salt water is placed into the front of the nose and then suctioned out. Poly-ICLC is then squirted into each nostril, one after the other, at a dose of 0.25, 0.5 or 1 mg. A small number of subjects are given a placebo (a solution with no active ingredient.) Subjects are observed in the clinic for 30 minutes after treatment.
* Day 2: Subjects receive a second nasal wash and repeat blood tests. They keep a diary card for 1 week, recording any drug side effects.
* Day 5: Subjects have repeat blood tests and a review of their diary card. The keep a diary card for another 3 weeks.
* Day 12: Subjects are contacted by phone to review their diary card.
* Day 28: Subjects are contacted by phone to review their diary card.

Part II

* Up to 7 days before Poly-ICLC administration: Medical history, physical examination and blood tests.
* Day 1: Nasal wash and Poly-ICLC administration. Same as above for Part I participants.
* Day 3: Subjects receive a second dose of medication and are observed again for 30 minutes.
* Day 4: Subjects receive a second nasal wash and repeat blood tests. They keep a diary card for 1 week, recording any drug side effects.
* Day 7: Subjects have repeat blood tests and a review of their diary card. The keep a diary card for another 3 weeks.
* Day 14: Subjects are contacted by phone to review their diary card.
* Day 28: Subjects are contacted by phone to review their diary card.

DETAILED DESCRIPTION:
Polyinosinic-Polycytidylic acid stabilized with polylysine and carboxymethylcellulose (Poly-ICLC), a stabilized double stranded RNA (dsRNA) therapeutic viral mimic activating innate and adaptive immunity, has been in extensive preclinical and investigational clinical therapeutic use as an intramuscular and intravenous compound, most recently in oncology applications. Only recently have the mechanisms of action been more fully elucidated, including induction of interferons, cytokines, and chemokines. Recognizing this, the infectious disease applications have been pursued in in vitro and animal models. Intranasal Poly-ICLC provides protection against mortality in animal models for multiple highly pathogenic viruses including influenza, severe acute respiratory distress syndrome (SARS), smallpox and Ebola. As its effects are not dependant on knowing the causative virus, an effective compound that could be protective against several unknown respiratory viruses has significant clinical appeal. While there is clinical safety data for intramuscular (IM) Poly-ICLC, no clinical studies of nasal application of Poly-ICLC have been done.

This study is a phase I safety and pharmacokinetic trial of nasally applied Poly-ICLC. Human volunteers will be administered increasing doses of nasal Poly-ICLC, with serial evaluation of safety, tolerability, as well as exploratory markers of immune activation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers age greater than or equal to 18 years and less than or equal to 70 years.

For 2 months prior to study drug administration, and through the last day of follow-up (Day 28), subjects must agree to:

* Not take any topical nasal medications (prescription or over the counter).
* Not receive live attenuated influenza vaccine (Flumist) or any other live attenuated intranasal vaccine (licensed or research).
* Not receive any other investigational medications or vaccines.

Females of child-bearing potential must agree to use one of the following methods of contraception for 4 weeks prior to date of screening evaluation through 4 weeks after study drug administration:

* Be surgically sterile.
* Use oral contraceptives or other form of hormonal birth control including hormonal vaginal rings or transdermal patches.
* Use an intra-uterine device (IUD).
* Use (by ensuring her male partner(s) uses) barrier contraception (condom) with a spermicide.
* Any other equivalent (as judged by the investigative team) methods of contraception.

EXCLUSION CRITERIA:

A medical history that includes any of the following:

Any chronic medical problem that requires daily topical nasal medications.

Prior nasal or sinus surgery (including trans-nasal approaches of other organs such as pituitary).

Allergic rhinitis, chronic sinusitis, or any other nasal inflammatory disease that requires daily intranasal or oral medication.

Any chronic pulmonary conditions including (but not limited to) asthma, chronic obstructive pulmonary disease, and chronic bronchitis.

Subjects with known hypersensitivity to interferons.

Any other medical history that in the opinion of the investigator significantly increases the risk associated with a Phase I drug (e.g. Patients with coronary heart disease, congestive heart failure, HIV, neuropsychiatric disorders, seizure disorder, autoimmune disease, hepatic decompensation, poorly controlled endocrine disorders (including poorly controlled diabetes, and actively hyper- or hypo-thyroid), hematological disorders (e.g. leukopenia, thrombocytopenia), ophthalmologic disorders (excluding errors or refractiveness) or other disorders for which symptoms of the condition could be similar to interferon-related toxicity or that might be exacerbated by interferon would be excluded. Patients with mild stable conditions, such as controlled hypertension, controlled diabetes, and osteoarthritis would be permitted to enroll.)

Any history of habitual intranasal cocaine or other intranasal recreational drug use at any time, or experimental intranasal concaine or other intranasal recreational drug use within the last 10 years. (e.g. a 50 year old who tried cocaine once at age 20 is acceptable for enrollment).

Women who are breast-feeding.

Positive urine or serum pregnancy test.

Participation in any research protocol that requires more than 100cc of blood to be given in any 6-week period of time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-03-24; Primary Completion 2009-12-16 (Actual); Study Completion 2009-12-16 (Actual)

PRIMARY OUTCOMES:
Frequency of AE greater than or equal to grade 2 by subjects who receive drug

SECONDARY OUTCOMES:
Intranasal cytokines, nasal NO production, inflammatory cells in nasal wash

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dushoff J, Plotkin JB, Viboud C, Earn DJ, Simonsen L. Mortality due to influenza in the United States--an annualized regression approach using multiple-cause mortality data. Am J Epidemiol. 2006 Jan 15;163(2):181-7. doi: 10.1093/aje/kwj024. Epub 2005 Nov 30. PMID 16319291
- [Background] Hui DS, Sung JJ. Severe acute respiratory syndrome. Chest. 2003 Jul;124(1):12-5. doi: 10.1378/chest.124.1.12. No abstract available. PMID 12853495
- [Background] Shortridge KF. Severe acute respiratory syndrome and influenza: virus incursions from southern China. Am J Respir Crit Care Med. 2003 Dec 15;168(12):1416-20. doi: 10.1164/rccm.2310005. No abstract available. PMID 14668255